CLINICAL TRIAL: NCT00467818
Title: Omega 3 Fatty Acids in the Treatment of Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sherie Novotny, M.D., Assistant Professor, Psychiatry, RWJMS, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220060238; 5R21AT002927 (NIH)
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Autism
Keywords: Aggression; Irritability; Global severity
MeSH Terms: conditions — Autistic Disorder; Aggression | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega 3 fatty Acids, drug (Active Comparator): Omega 3 Fatty acids will be dispensed to subjects in the active experimental group of the study.
  Interventions: Drug: Omega 3 fatty acids
- Placebo (Placebo Comparator): The placebo will be dispensed to subjects in the control group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omega 3 fatty acids — The study will start with low doses and based on the weight of the individual the dosage will be increased biweekly.
  Other Names: DHA and EPA
  Arms: Omega 3 fatty Acids, drug
Other: Placebo — Same dosage as that of omega 3 fatty acids
  Arms: Placebo

SUMMARY:
Published studies on omega 3 fatty acids in the treatment of bipolar disorder and schizophrenia have shown reductions in time to recurrence, a decrease in the positive and negative symptoms of schizophrenia, and improvements in Clinical Global Impression Scale, Young Mania Rating Scale, and HAM-D scores. The following are the hypotheses:

* Omega 3 fatty acids will be superior to placebo in the acute treatment of global autism.
* Omega 3 fatty acids will be superior to placebo in improving aggression and irritability associated with autism.
* Omega 3 fatty acids will be superior to placebo in improving functional ability.

DETAILED DESCRIPTION:
This study is an innovative treatment approach to autism. It adapts a promising adjunct therapy for bipolar disorder and schizophrenia to a new population, that of children and adolescents with autism. It will analyze the possible relationship between dosage of omega 3 fatty acids and treatment outcomes. Finally, it will attempt to identify which specific subgroups of subjects will respond to this intervention, which components and associated features are most responsive and whether this impacts subjects' quality of life. The data generated by this study is intended to support the rationale for a full scale, large multi-site clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Child/Teen has autism.
* He/She is between five and seventeen years of age.
* He/She is not in the hospital.
* He/She has a parent or legal guardian who is willing and able to sign the informed consent.

Exclusion Criteria:

* Child/Teen has been diagnosed with a psychotic disorder (such as schizophrenia) or a mood disorder, including depression or bipolar disorder (manic depression).
* He/She has caused visible harm to him/herself or is at risk for suicide.
* He/She has an active seizure disorder or epilepsy (seizures within the past year).
* He/She has an unstable medical illness, including heart disease.
* He/She has experienced brain injury.
* He/She has a history of diabetes.
* He/She has a history of prior treatment with Omega 3 Fatty Acids.
* He/She lives in a far away area and/or does not have regular access to transportation to the clinical facility.
* A pregnant female or unwilling to use acceptable contraception if sexually active.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherie L. Novotny, MD, Principal Investigator — Division of Child and Adolescent Psychiatry at the University of Medicine and Dentistry of New Jersey
Locations (1):
- University Behavioral Health Care Building, UMDNJ-RWJMS, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time.

REFERENCES:
- [Result] Amminger GP, Berger GE, Schafer MR, Klier C, Friedrich MH, Feucht M. Omega-3 Fatty Acids Supplementation in Children with Autism. Biol Psychiatry. 2006 Aug 22 Harel Z, Gascon G, Riggs S, Vaz R, Brown W, Exil G. Supplementation with omega-3 polyunsaturated fatty acids in the management of recurrent migraines in adolescents. J Adolesc Health. 2002 Aug;31(2):154-61. Itomura M, Hamazaki K, Sawazaki S, Kobayashi M, Terasawa K, Watanabe S, Hamazaki T. The effect of fish oil on physical aggression in schoolchildren. J Nutr Biochem. 2005 Mar;16(3):163-71. Mitchell EA, Aman MG, Turbott SH, Manku M. Clinical characteristics and serum essential fatty acid levels in hyperactive children. Clin Pediatr 1987; 26:406-11. Nemets H, Nemets B, Apter A, Bracha Z, Belmaker RH Omega-3 treatment of childhood depression: Am J Psychiatry. 2006 Jun;163(6):1098-100. Richardson AJ, Montgomery P. The Oxford-Durham study. Pediatrics. 2005 May;115(5):1360-6.
- See also: University Behavior Health Care official website — http://ubhc.umdnj.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was difficult for this study due to multiple disruptions in the flow of the study due to issues with the IRB process. Additionally, there were periods of time when there was not a research coordinator to assist with recruitment and pt flow.
Pre-assignment Details: Participants were required to undergo diagnostic testing and intelligence testing prior to starting the study. Individuals who were unable to participate in these processes were not allowed to enter into the active phase of the study.
Groups:
- Omega 3 Fatty Acids, Drug: Omega 3 Fatty acids will be dispensed to subjects in the active experimental group of the study.
  Omega 3 fatty acids : The study will start with low doses and based on the weight of the individual the dosage will be increased biweekly.
- Placebo: The placebo will be dispensed to subjects in the control group
  Placebo : Same dosage as that of omega 3 fatty acids
Period: Overall Study
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Started | 9 | 8
Completed | 6 | 6
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 8 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (3.5) | 10.6 (3.5) | 11.2 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale(CGI)- Improvement
Description: This scale measures the impression of improvement as assessed from interviewing the subject and informant.The scale is measured with numbers from 0 through 7 with 0 not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. Units = scores on a scale.
Time Frame: Administered biweekly, endpoint score (week 12) only used for data analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 3.57 (1.2) | 3.8 (1.2)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids, Drug vs Placebo; Test type: Superiority or Other; p = 1.0, t-test, 2 sided

2. Primary Outcome: Aberrant Behavior Checklist (ABC)
Description: Aberrant Behavior Checklist (ABC)-Community Version (Irritability Subscale) (Aman et al. 1985). It is designed to objectively identify five behavior subscales through observation by the primary caregiver. The five behavior subscales include (ranges show no problem to severe problem): irritability (range 0-45), lethargy (range 0-48), stereotypy (range 0-21), hyperactivity range 0-48), and inappropriate speech (range 0-12), all possible signs and symptoms of affective instability in autistic individuals (Lainhart & Folstein, 1994). Improvement is shown with scores decreasing over time. Total score is not used. Inter-rater reliability for the ABC-CV is moderate to high across subscales with a mean of .63. Test-retest reliability correlations are .98 -Irritability, .99 -Lethargy, .98 -Stereotypy, .98 -Hyperactivity, and .96 -Inappropriate Speech. The ABC will be filled out by an informant (teacher/parent), and then reviewed by the IE. Administration time is approximately 10 minutes.
Time Frame: Administered every 4 weeks, 12 week scores used for means, score on irritability subscale reported
Population: Youth and adolescents ages 5-17 with autism spectrum disorder
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 5.66 (5.0) | 8.5 (2.1)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids, Drug vs Placebo; Test type: Superiority; p = 0.10, Mixed Models Analysis; Mean Difference (Final Values) = 0.10

3. Primary Outcome: Vineland Adaptive Behavior Scale
Description: The Vineland Scale is a semi-structured informant interview that assesses subjects' functioning. It is administered to a caretaker/family member. The scale has been revised and standardized in all populations. This scale has been found to assess social deficits in autism and strengths in daily living skills. Items are classified under four major adaptive domains: communication, daily living skills, socialization and motor skills. The items are scored 0-2 (yes/sometimes/never). Each domain is summed, and the domain scores are converted to standardized scores. The normative score is 100, with standard deviation of 15. The standardized score is used in this study. A higher score (above 100) means better adaptive behavior. Minimum value is 0, maximum value is infinity.
Time Frame: Administered during the baseline visit and on week 12 ( termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 51.5 (13.28) | 27.5 (9.81)

4. Secondary Outcome: Overt Aggression Scale-Modified
Description: The Modified version, Coccaro et al. is designed for outpatient use and assessment of behavior over one week. This scale was assessed biweekly. The OAS-M consists of 3 domains: Aggression, Irritability, and Suicidality (not used). Aggression Domain: 4 subscales of weighted behavior: Verbal Aggression (1), Aggression Against Objects (2), Aggression Against Others (3), and Self-Aggression (4). Within each category, severity of an event receives a scaled score (0-5) (higher score for worse behaviors) which is then multiplied by the weekly frequency of this event and weight, then totaled (for use in this study). Irritability subscale is divided into subjective/objective, 0 (low)-5 (high). The total scale has a minimum value of 0 (no display of aggressive/irritable behavior) and a maximum value of infinity (worse aggressive/irritable behavior) as reporting the number of times an aggressive/irritable behavior occurred does not have a maximum value). Higher scores mean worse outcome.
Time Frame: Administered biweekly and at week 12 (termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 3.8 (2.7) | 2.4 (2.6)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids, Drug vs Placebo; Test type: Superiority; p < 0.5, Mixed Models Analysis; Mean Difference (Final Values) = 0.50

5. Secondary Outcome: Parental Stress Index
Description: This measurement assesses child and parental characteristics and parent-child relationship dimensions associated with the presence of parenting stress/ troubled relationships. It is a self-report scale completed by the parent, consisting of 101 items organized into two domains with the following subscales: (1) child characteristics domain - adaptability, demandingness, mood, distractibility/hyperactivity, acceptability of child to parent, and child's reinforcement of parent, and (2) parent characteristics domain - depression, attachment to child, social isolation, sense of competence in the parenting role, relationship with spouse/parenting partner, role restrictions, and parental health. Scores are 1-5 with 1 being strongly agree and 5 being strongly disagree. Scores are collected and standardized. The higher a score is, the more stress a parent is experiencing. Minimum value is 101 and maximum value is 505.
Time Frame: Administered during the baseline visit and on week 12 ( termination)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 314.2 (35.2) | 279.5 (35.4)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acids, Drug vs Placebo; Test type: Superiority; p = 0.5, Mixed Models Analysis; Mean Difference (Final Values) = 0.5

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the course of the study from the start in 2007 until completion in 2011. Each participant was observed for adverse events during the course of their treatment which was the course of the study, ie 12 weeks. Participants were not monitored for adverse events after the completion of the study.
Arm/Group | Omega 3 Fatty Acids, Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega 3 Fatty Acids, Drug (N=9) | Placebo (N=8)
Recurrence of mood disorder in one participant (Psychiatric disorders) | 0 (0) | 1 (1) — One subject had a recurrence of a psychiatric issue ( although might be unrelated to the intake of the placebo which he was on) which lead to hospitalization and discontinuation of taking the placebo and subsequent withdrawal from the study.

LIMITATIONS AND CAVEATS:
One subject had a recurrence of a psychiatric issue ( although might be unrelated to the intake of the placebo which he was on) which lead to hospitalisation and discontinuation of taking the placebo and subsequent withdrawal from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No